CLINICAL TRIAL: NCT01779999
Title: Observational Study With Ultrasonographic Screening for Early Detection of PICC-related DVT, Results of Early Beginning of Anticoagulant Treatment
Brief Title: Early Detection of PICC-related Deep Vein Thrombosis by US Surveillance: an Effective Approach for Secondary Prevention?
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Cristina Garrino, PhD, University of Turin, Italy
Other Study IDs: SGB0012226
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Central Venous Catheter Thrombosis
Keywords: central venous catheters; thrombosis; secondary prevention
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PICC-carrying patients: All patients carrying a peripherally inserted central catheter in our service
  Interventions: Other: PICC-carrying patients

INTERVENTIONS:
Other: PICC-carrying patients — Echographic monitoring of patients carrying a peripherally inserted central catheter

SUMMARY:
Background: PICC-related thrombosis have shown a slightly different pattern of frequency and risk factors, compared with traditional CVC; because of the increasing diffusion of PICCs, they are becoming a somehow independent pathology, still under investigation; no pharmacological prevention has proved to be effective. Aim of this study is to estimate the cumulative incidence of thrombosis in a cohort of patients carrying a PICC-line CVC, monitored to allow an early detection and prevention of complications related to the presence of asymptomatic deep venous thrombosis, and to explore the role of several potential risk factors.

Methods: in a prospective observational cohort we will enroll 150 consecutive patients having a PICC inserted by our team; clinical characteristics, comorbidities and main features of catheter positioning procedure will be registered; patients will be followed with clinical and echographic scheduled controls, weekly for the first month, then monthly; patients with PRDVT will be treated with LMWH and recontrolled weekly until removal of catheter

DETAILED DESCRIPTION:
All PICCs are positioned by trained physicians and nurses, after ultrasonographic screening of the whole upper limbs venous district, axillary, subclavian and jugular veins for detecting possible pre-existing thrombosis; positioning is performed with real-time ultrasonography guide with a portable device. Patients are recontrolled one week after positioning; patients who report pain, swelling, fever, skin colour changes, exit site tenderness, or any symptom suspected for thrombosis or infection, are immediately seen. A duplex ultrasound complete examination of the upper limb and neck vessels is performed, and at the same time the whole arm and the exit site is inspected to exclude infections; diagnostic criteria for DVT include incompressibility of the vein and direct visualisation of PICC-surrounding thrombus; in uncertain cases, a doppler examination is performed.If the examination is negative for thrombosis, further controls are performed at 2,3,4 weeks after positioning, then once a month.If a DVT is detected, we register the position and extension of the thrombus, and its main characteristics (clot, mural or occlusive thrombosis); the catheter is left in place and a therapy is prescribed with LMWH at full doses, according with ACCP guidelines 2008 (confirmed in 2012 edition). Then, the patient is recontrolled weekly until removal of the catheter.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a PICC-line positioning during a five-months period

Exclusion Criteria:

* age<18,complete paresis of the arm, history of previous DVT in the same arm, expected very short PICC indwelling time (less than 1 week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a PICC-line positioning during a five-months period
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
early detection of PRDVT | 1 yr
  weekly ultrasonographic examination of the whole upper limbs venous district, axillary, subclavian and jugular veins for detecting incompressibility of the vein or visualization of thrombus; Doppler examination for confirmation of DVT

SECONDARY OUTCOMES:
risk factors individuation | 1 yr

OTHER OUTCOMES:
DVT resolution with early therapy | 1yr

CONTACTS AND LOCATIONS:
Overall Officials: cristina garrino, PhD, Principal Investigator — University of Turin, Italy